CLINICAL TRIAL: NCT02744105
Title: Effect of Spirulina on Liver Fibrosis by Transient Elastography in Beta Thalassemic Children With Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Elshanshory, head of pediatric hematology and oncology unit, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2902/11/14
Record Dates: First submitted 2016-04-16; First posted 2016-04-20 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- thalassemic children with hepatitis C (Experimental): 30 multitransfused beta thalassemic children infected with hepatitis C virus diagnosed by serological detection of HCV-antibodies and HCV RNA by polymerase chain reaction will be given Spirulina in a dose of 250 mg/kg/day orally for 3 months.
  Interventions: Dietary Supplement: Spirulina
- thalassemic children without hepatitis C (No Intervention): 30 multitransfused beta thalassemic children without hepatitis C virus infection

INTERVENTIONS:
Dietary Supplement: Spirulina — Spirulina in a dose of 250 mg/kg/day will be given orally for 3 months.
  Arms: thalassemic children with hepatitis C

SUMMARY:
Thalassemics can develop liver fibrosis because of iron overload and hepatitis C infection. The latter is the main risk factor for liver fibrosis in transfusion dependent thalassemics. Excess liver iron is clearly recognized as a co factor for the development of advanced fibrosis in patients with hepatitis virus C infection. Transient elastography (Fibroscan) is a reliable non invasive method for diagnosing as liver fibrosis in thalassemic patients regardless of the degree of iron overload. There is evidence that suggests Spirulina may help to protect against liver damage, cirrhosis and liver failure in those with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* multitransfused beta thalassemic children with and without super added hepatitis C virus (HCV) infection diagnosed by serological detection of HCV antibodies and HCV RNA by polymerase chain reaction.

Exclusion Criteria:

* liver decompensation child younger than 3 years patients with hepatitis B infection implantable cardiac device failure to obtain transient elastography (Fibroscan) results

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
liver stiffness measurement using transient elastography (Fibroscan) | 3 months

SECONDARY OUTCOMES:
liver function tests | 3 months
aspartate aminotransferase to platelet ratio index (APRI) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt